CLINICAL TRIAL: NCT02288117
Title: Prospective Clinical 5-year Follow-up of the LINK® SP-CL® Hip Prosthesis Stem
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Waldemar Link GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: 1202 HP
Record Dates: First submitted 2014-11-06; First posted 2014-11-11 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Osteoarthritis, Hip; Femur Head Necrosis; Femoral Neck Fractures
Keywords: PMCF; Post Market Clinical Follow up; SP-CL; anatomic stem
MeSH Terms: conditions — Osteoarthritis, Hip; Femur Head Necrosis; Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this PMCF is to collect clinical and radiographic outcome information on Total Hip Arthroplasty (THA) performed with LINK® SP-CL® Hip Prosthesis Stem under routine conditions.

The results collected will be used to clinically confirm the performance and safety of the LINK® SP-CL® Hip Prosthesis Stem in terms of the manufacturer's obligation to perform a PMCF. Furthermore the results can be used for future regulatory processes if needed.

DETAILED DESCRIPTION:
Post Market Clinical Follow-ups (PMCF) through observational studies are an important tool to detect infrequent complications or problems, events specific to defined patient populations and long term performance issues under routine conditions [2,3]. Against this background a prospective multi-center outcome study of the LINK® SP-CL® is planned.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature
* Subject agrees to comply with the required postoperative management and follow-up evaluations
* Undergone at least six (6) month of unsuccessful, conservative, non-surgical treatment
* Patient understands the conditions of the study and is willing and able to comply with the postoperative scheduled clinical and radiographic evaluations and the prescribed postoperative management.
* Patient signed Informed Consent.

Exclusion Criteria:

* Body Mass Index (BMI) > 40 kg/m2
* Poor general state of health
* Acute and chronic infections, local and systemic
* Pharmaceutical or other drug abuse, alcoholism
* Allergies to implant materials
* Distinctive muscular, nerve, vascular or other diseases which put the affected limb at risk
* Insufficient / inadequate bone mass- or quality which prevents a stable anchorage of the prosthesis
* Severe osteoporosis
* Foreseeable overload/ overstressing of the joint prosthesis
* Acetabular defects
* Female patient who is pregnant or plans to became pregnant during the course of the study
* Prisoner
* Patient who, as judged by the surgeon, is mentally incompetent or is unlikely to be compliant with the prescribed postoperative routine and follow-up evaluation schedule
* Patient who has not signed the Informed Consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mobility-limiting disease, fracture or defect of the hip joint requiring primary THA with SP-CL® (i.e. primary or secondary coxarthrosis, osteoarthritis, femoral neck fracture, necrosis of the femoral head)
  ·
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Stem Survival Rate | Up to 5 years
  The survival of the stem

SECONDARY OUTCOMES:
Complication Rate | Up to 5 years
  Number and kind of complications
Reoperation Rate | Up to 5 years
  number of reoperations
Harris Hip Score (HHS) | Up to 5 years
  Clinical Score to get information about the subjects pain and hip function, collected continuously
Oxford Hip Score (OHS) | Up to 5 years
  PROM to assess function and pain after THR
Forgotten Joint Score (FJS) | Up to 2 years
  awareness of the artificial joint
Mid Thigh Pain | Up to 5 years
  Pain occuring in the front and mid part of the femur

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Gehrke, Prof. Dr., Principal Investigator — HELIOS Endo-Klinik Hamburg
Locations (4):
- Germany (2):
  - Krankenhaus Barmherzige Brüder Regensburg, Regensburg, Bavaria
  - HELIOS ENDO-Klinik, Hamburg
- L'Istituto Ortopedico Gaetano Pini, Milan, Italy
- Hospital Sant Rafael, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided